CLINICAL TRIAL: NCT01950728
Title: Hypoalgesic Effect of Low Frequency and Burst Modulated Alternating Currents on Healthy Individuals.
Brief Title: Electrical Currents on Hypoalgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fabio Massao Matuzawa (Other)
Responsible Party: Sponsor-Investigator, Fabio Massao Matuzawa, Physical Therapy Student, Paulista University
Organization: Paulista University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14571013.1.0000.5512
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: volunteers; 18 to 65 years; Males and Females
MeSH Terms: interventions — Electric Stimulation Therapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): This group will not receive electrical stimulation. Volunteers will rest during 30 minutes.
- Interferential current group (Active Comparator): Interferential current will be applied during 30 minutes to volunteer's forearm. Intensity will be increase until volunteers fell a strong but comfortable paresthesia.
  Interventions: Device: Interferential current
- TENS Group (Active Comparator): TENS will be applied during 30 minutes to volunteer's forearm. Intensity will be increase until volunteers fell a strong but comfortable paresthesia.
  Interventions: Device: TENS
- Aussie current group (Active Comparator): Aussie current will be applied during 30 minutes to volunteer's forearm. Intensity will be increase until volunteers fell a strong but comfortable paresthesia.
  Interventions: Device: Aussie Current

INTERVENTIONS:
Device: Interferential current — Interferential current will be applied during 30 minutes to volunteer's forearm at a strong but comfortable intensity. Carrier frequency will be set at 4 kilohertz (kHz) and modulated frequency will be set at 100 Hz.
  Arms: Interferential current group
Device: Aussie Current — Aussie current will be applied during 30 minutes to volunteer's forearm at a strong but comfortable intensity. Carrier frequency will be set at 4 kHz and modulated frequency will be set at 100 Hz.
  Arms: Aussie current group
Device: TENS — TENS will be applied during 30 minutes to volunteer's forearm at a strong but comfortable intensity. Pulse duration will be set at 125 microseconds and frequency will be set at 100 Hz.
  Arms: TENS Group

SUMMARY:
The objective of this study is to compare the hypoalgesic effects of TENS, Interferential current and Aussie current in pressure pain threshold and sensory discomfort in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* health adults

Exclusion Criteria:

* injury to nerves of the upper limbs, pain, pregnancy, chronic diseases, cardiac pacemaker, epilepsy, allergy to the electrode used, use of pain medication, skin lesions or lack of sensitivity in the areas of electrode placement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2018-01-23 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold | Baseline, 15 minutes after the beginning of electrical stimulation, 30 minutes after the beginning of electrical stimulation, and 20 minutes after electrical stimulation.
  Pressure Pain Threshold will be measured using a digital pressure algometer SOMEDIC type II. The applied force will be measured in Newton (N).

SECONDARY OUTCOMES:
Sensory Discomfort | 15 and 30 minutes after the beginning of electrical stimulation.
  Sensory Discomfort will be measured using a 10 cm visual analogue scale (VAS). The degree of discomfort will be measured in centimeters (cm).

CONTACTS AND LOCATIONS:
Locations (1):
- CPA Pompéia UNIP, São Paulo, Brazil

REFERENCES:
- [Derived] Rampazo da Silva EP, da Silva VR, Bernardes AS, Matuzawa FM, Liebano RE. Study protocol of hypoalgesic effects of low frequency and burst-modulated alternating currents on healthy individuals. Pain Manag. 2018 Mar;8(2):71-77. doi: 10.2217/pmt-2017-0058. Epub 2018 Feb 16. PMID 29451431